CLINICAL TRIAL: NCT03645330
Title: Prospective Multicenter Observational Study of Atezolizumab in Patients With Unresectable, Locally Advanced or Metastatic Non-small Cell Lung Cancer: (J-TAIL)
Brief Title: A Study of Atezolizumab in Patients With Unresectable, Locally Advanced or Metastatic NSCLC (J-TAIL)
Status: Completed | Type: Observational
Sponsor: Chugai Pharmaceutical (Industry)
Collaborators: Japan Lung Cancer Society (Other)
Responsible Party: Sponsor
Other Study IDs: J-TAIL
Record Dates: First submitted 2018-08-19; First posted 2018-08-24 (Actual); Last update posted 2022-07-22 (Actual); Status verified 2022-07

CONDITIONS: Non-small-Cell Lung Cancer
Keywords: Atezolizumab
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This prospective, observational study is to assess the long-term effectiveness and safety of Atezolizumab in patients with advanced non-small cell lung cancer in clinical practice.

DETAILED DESCRIPTION:
Primary endpoint: 18 months OS, Secondary endpoints: Overall Survival(OS), 12 months survival rate(12mo OS), 24 months survival rate(24mo OS), Progression-Free Survival(PFS), Time to treatment failure (TTF), Objective Response Rate(ORR), Disease Control Rate(DCR), Duration of Response(DOR) ,Safety and EuroQol 5-Dimension 5-Level (EQ-5D-5L) Questionnaire

ELIGIBILITY:
Inclusion Criteria:

* Patients 20 years of age or older at the time of signed consent.
* Patients with locally advanced or metastatic non-small cell lung cancer.
* Patients who are scheduled to start Atezolizumab monotherapy, based on the Atezolizumab package insert and the Optimal Use Promotion Guideline.
* Patients who signed informed consent form before enrolling the study. The consent from a legally acceptable representative is required for the patients with uncertain capacity of judgments.

Exclusion Criteria:

* Patients who are considered to be unsuitable for enrolment into the study by the investigator's judgment.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are planning to provide Atezolizumab monotherapy as the most appropriate medical care for patients and who meet the Eligibility criteria at registration.
Sampling Method: Probability Sample
Enrollment: 1026 (Actual)
Dates: Start 2018-08-15 (Actual); Primary Completion 2021-07-08 (Actual); Study Completion 2021-07-08 (Actual)

PRIMARY OUTCOMES:
18 months survival rate | Baseline up to 18 Months
  Percentage of participants alive 18 months after initiation of treatment

SECONDARY OUTCOMES:
Overall Survival(OS) | Up to death (up to 4 years)
  OS was defined as the time from the first day of study treatment to death due to any cause
12 months survival rate | Up to 12 months
  Percentage of participants alive 12 months after initiation of treatment
24 months survival rate | Up to 24 months
  Percentage of participants alive 24 months after initiation of treatment
Progression-Free Survival(PFS) | Up to disease progression or death whichever occurs first (up to 4 years)
  PFS based on disease status as evaluated by the investigator in accordance with Response Evaluation Criteria in Solid Tumors (RECIST), Version 1.1 (v1.1)
Time to treatment failure (TTF) | Up to 4 years
  TTF was defined as the time from the first day of study treatment to treatment discontinuation for any reason, including disease progression, treatment toxicity, patient preference, or death
Objective Response Rate(ORR) | Up to disease progression or death whichever occurs first (up to 4 years)
  Percentage of participants with objective response as assessed by the investigator according to RECIST v1.1
Disease Control Rate(DCR) | Up to 4 years
  Percentage of patients with controled disease as Assessed by the investigator according to RECIST v1.1
Duration of Response(DOR) | From date of first objective response up to disease progression or death whichever occurs first (up to 4 years)
  Duration of Response as Assessed by the Investigator According to RECIST v1.1
Percentage of Participants with adverse events(Adverse Reactions) | Up to 4 years
  The incidence of worst-grade adverse events on study as graded by NCI-CTCAE v4.0
EuroQol 5-Dimension 5-Level (EQ-5D-5L) Questionnaire | Day 1 of first cycle(21-day cycle), then every 12 weeks until disease progression or until treatment discontinuation(Up to 4 years)
  EQ-5D-5L consists of five standardized questions. Evaluate the quality of life by converting the result obtained into scores (range: 1.000 to - 0.025). Higher values give better results.

CONTACTS AND LOCATIONS:
Overall Officials: Tetsuya MITSUDOMI, MD/PhD, Principal Investigator — Kindai University Faculty of Medicine
Locations (198):
- Japan (198):
  - Akashi Medical Center, Akashi
  - Hyogo Cancer Center, Akashi
  - Akita University Hospital, Akita
  - Hyogo Prefectural Amagasaki General Medical Center, Amagasaki
  - Aomori Prefectural Central Hospital, Aomori
  - Asahikawa Medical University Hospital, Asahikawa
  - National Hospital Organization Asahikawa Medical Center, Asahikawa
  - Juntendo University Hospital, Bunkyō City
  - Nippon Medical School Hospital, Bunkyō City
  - Tokyo Medical And Dental University, Medical Hospital, Bunkyō City
  - Tokyo Metropolitan Cancer and Infectious disease Center Komagome Hospital, Bunkyō City
  - Chiba Cancer Center, Chiba
  - Chiba University Hospital, Chiba
  - National Cancer Center Hospital, Chūōku
  - Fujisawa City Hospital, Fujisawa
  - Fukui Prefectural Hospital, Fukui
  - Fukuoka University Hospital, Fukuoka
  - Kyushu University Hospital, Fukuoka
  - National Hospital Organization Kyushu Cancer Center, Fukuoka
  - National Hospital Organization Kyushu Medical Center, Fukuoka
  - Fukushima Medical University Hospital, Fukushima
  - Funabashi Municipal Medical Center, Funabashi
  - Gifu Prefectural General Medical Center, Gifu
  - Gifu University Hospital, Gifu
  - National Hospital Organization Okinawa National Hospital, Ginowan
  - Osaka Habikino Medical Center, Habikino
  - Hamamatsu University Hospital, Hamamatsu
  - National Hospital Organization Himeji Medical Center, Himeji
  - Hirosaki University Hospital, Hirosaki
  - National Hospital Organization Hirosaki National Hospital, Hirosaki
  - Hiroshima City Hiroshima Citizens Hospital, Hiroshima
  - Hiroshima Prefectural Hospital, Hiroshima
  - Hiroshima University Hospital, Hiroshima
  - Tokyo Medical University Ibaraki Medical Center, Ibaraki
  - Iizuka Hospital, Iizuka
  - Nippon Medical School Chiba Hokusoh Hospital, Inzai
  - Japanese Red Cross Ise Hospital, Ise
  - Tokai University Hospital, Isehara
  - Isesaki Municipal Hospital, Isesaki
  - Itami City Hospital, Itami
  - National Hospital Organization Iwakuni Clinical Center, Iwakuni
  - Shimane University Hospital, Izumo
  - Juntendo University Shizuoka Hospital, Izunokuni
  - Kagawa University Hospital, Kagawa
  - Kagoshima University Hospital, Kagoshima
  - Kameda Medical Center, Kamogawa
  - Ishikawa Prefectural Central Hospital, Kanazawa
  - Kanazawa University Hospital, Kanazawa
  - Ibaraki Prefectural Central Hospital, Kasama
  - Kasukabe Medical Center, Kasukabe
  - Kanto Rosai Hospital, Kawasaki
  - Kawasaki Municipal Hospital, Kawasaki
  - Kimitsu Chuo Hospital, Kisarazu
  - Kishiwada City Hospital, Kishiwada
  - Hospital of the University of Occupational and Envioronmental Health, Japan, Kitakyushu
  - Japan Community Health care Organization Kyushu Hospital, Kitakyushu
  - Kitakyushu Municipal Medical Center, Kitakyushu
  - Fukujuji Hospital, Kiyose
  - National Hospital Organization Tokyo National Hospital, Kiyose
  - Kobe City Medical Center General Hospital, Kobe
  - Kobe Minimally Invasive Cancer Center, Kobe
  - Kobe University Hospital, Kobe
  - Yamanashi Prefectural Central Hospital, Kofu
  - Komatsu Municipal Hospital, Komatsu
  - Dokkyo Medical University Saitama Medical Center, Koshigaya
  - Ohta Nishinouchi Hospital, Kōriyama
  - Cancer Institute Hospital of Japanese Foundation For Cancer Research, Kōtoku
  - Kumamoto Regional Medical Center, Kumamoto
  - Kumamoto University Hospital, Kumamoto
  - Kurashiki Central Hospital, Kurashiki
  - National Hospital Organization Kure Medical Center and Chugoku Cancer Center, Kure
  - Kurume University Hospital, Kurume
  - Japanese Red Cross Kyoto Daiichi Hospital, Kyoto
  - Japanese Red Cross Kyoto Daini Hospital, Kyoto
  - Kyoto City Hospital, Kyoto
  - Kyoto University Hospital, Kyoto
  - Kyoto-Katsura Hospital, Kyoto
  - National Hospital Organization Kyoto Medical Center, Kyoto
  - University Hospital, Kyoto Prefectural University of Medicine, Kyoto
  - Gunma University Hospital, Maebashi
  - Shinshu University Hospital, Matsumoto
  - Matsusaka Municipal Hospital, Matsusaka
  - Ehime Prefectural Central Hospital, Matsuyama
  - Matsuyama Red Cross Hospital, Matsuyama
  - National Hospital Organization Shikoku Cancer Center, Matsuyama
  - National Hospital Organization Tokyo Medical Center, Meguro City
  - The Jikei University Hospital, Minatoku
  - Tokyo Saiseikai Central Hospital, Minatoku
  - Toranomon Hospital, Minatoku
  - Kyorin University Hospital, Mitaka
  - Miyazaki Prefectural Miyazaki Hospital, Miyazaki
  - Iwate Prefectural Central Hospital, Morioka
  - Shiga General Hospital, Moriyama
  - Nagahama City Hospital, Nagahama
  - Aichi Medical University Hospital, Nagakute
  - Japanese Red Cross Society Nagano Hospital, Nagano
  - Nagaoka Red Cross Hospital, Nagaoka
  - Nagasaki University Hospital, Nagasaki
  - Aichi Cancer Center, Nagoya
  - Japanese Red Cross Nagoya Daini Hospital, Nagoya
  - Nagoya City West Medical Center, Nagoya
  - Nagoya Ekisaikai Hospital, Nagoya
  - Nagoya University Hospital, Nagoya
  - National Hospital Organization Nagoya Medical Center, Nagoya
  - Kochi Medical School Hospital, Nankoku
  - Nara Prefecture General Medical Center, Nara
  - Miyagi Cancer Center, Natori
  - Niigata Cancer Center Hospital, Niigata
  - Niigata University Medical and Dental Hospital, Niigata
  - The Hospital of Hyogo College of Medicine, Nishinomiya
  - Obihiro Kosei Hospital, Obihiro
  - Japanese Red Cross Okayama Hospital, Okayama
  - Kawasaki Medical School General Medical Center, Okayama
  - Okayama Rosai Hospital, Okayama
  - Okayama University Hospital, Okayama
  - University of Ryukyus Hospital, Okinawa
  - Kitano Hospital, Osaka
  - Osaka City General Hospital, Osaka
  - Osaka City University Hospital, Osaka
  - Osaka General Medical Center, Osaka
  - Osaka International Cancer Institute, Osaka
  - Osaka Medical College Hospital, Osaka
  - Osaka Police Hospital, Osaka
  - Osaka Red Cross Hospital, Osaka
  - Osaka Saiseikai Nakatsu Hospital, Osaka
  - Ogaki Municipal Hospital, Ōgaki
  - Oita Prefectural Hospital, Ōita
  - Kindai University Hospital, Ōsaka-sayama
  - Osaki Citizen Hospital, Ōsaki
  - Gunma Prefectural Cancer Center, Ōta-ku
  - Shiga University of Medical Science Hospital, Ōtsu
  - Saga University Hospital, Saga
  - Kitasato University Hospital, Sagamihara
  - Jichi Medical University Saitama Medical Center, Saitama
  - Saitama Cancer Center, Saitama
  - Saitama Medical University Hospital, Saitama
  - Saitama medical university International medical Center, Saitama
  - Saitama Red Cross Hospital, Saitama
  - National Hospital Organization Kinki-Chuo Chest Medical Center, Sakai
  - Nihonkai General Hospital, Sakata
  - Hokkaido Cancer Center, Sapporo
  - Hokkaido University Hospital, Sapporo
  - Japan Community Health care Organization Hokkaido Hospital, Sapporo
  - Sapporo Medical University Hospital, Sapporo
  - Teine Keijinkai Hospital, Sapporo
  - Sendai Medical Association Hospital, Sendai
  - Sendai Kousei Hospital, Sendai
  - Tohoku Medical And Pharmaceutical University Hospital, Sendai
  - Tohoku University Hospital, Sendai
  - Tosei General Hospital, Seto
  - Japanese Red Cross Medical Center, Shibuya City
  - Jichi Medical University Hospital, Shimotsuke
  - NTT Medical Center Tokyo, Shinagawa-Ku
  - Showa University Hospital, Shinagawa-Ku
  - Center Hospital of the National Center for Global, Shinjuku-Ku
  - Keio University Hospital, Shinjuku-Ku
  - Tokyo Medical University Hospital, Shinjuku-Ku
  - Tokyo Women's Medical University Hospital, Shinjuku-Ku
  - Iwate Medical University Hospital, Shiwa-gun
  - Shizuoka Cancer Center, Shizuoka
  - Shizuoka General Hospital, Shizuoka
  - Osaka University Hospital, Suita
  - Saiseikai Suita Hospital, Suita
  - Gifu Prefectural Tajimi Hospital, Tajimi
  - Kagawa Prefectural Central Hospital, Takamatsu
  - KKR Takamatsu Hospital, Takamatsu
  - JA Toyama Kouseiren Takaoka Hospital, Takaoka
  - Takarazuka City Hospital, Takarazuka
  - Tenri Hospital, Tenri
  - Dokkyo Medical University Hospital, Tochigi
  - Tokushima Prefectural Central Hospital, Tokushima
  - Tokushima University Hospital, Tokushima
  - Toyama Prefectural Central Hospital, Toyama
  - Fujita Health University Hospital, Toyoake
  - Toyohashi Municipal Hospital, Toyohashi
  - Osaka Toneyama Medical Center, Toyonaka
  - TOYOTA Memorial Hospital, Toyota
  - Ehime University Hospital, Tōon
  - Mie University Hospital, Tsu
  - Tsukuba Medical Center Foundation, Tsukuba
  - University of Tsukuba Hospital, Tsukuba
  - National Hospital Organization Yamaguchi-Ube Medical Center, Ube
  - Uji-TOKUSHUKAI MEDICAL CENTER, Uji
  - Juntendo University Urayasu Hospital, Urayasu
  - Saiseikai Utsunomiya Hospital, Utsunomiya
  - Tochigi Cancer Center, Utsunomiya
  - Japanese Red Cross Wakayama Medical Center, Wakayama
  - Wakayama Medical University Hospital, Wakayama
  - Yamagata University Hospital, Yamagata
  - Yamaguchi University Hospital, Yamaguchi
  - Kanagawa Cancer Center, Yokohama
  - Kanagawa Cardiovascular and Respiratory Center, Yokohama
  - Yokohama City University Hospital, Yokohama
  - Yokohama City University Medical Center, Yokohama
  - Yokohama Municipal Citizen's Hospital, Yokohama
  - Yokosuka Kyosai Hospital, Yokosuka
  - Tottori University Hospital, Yonago
  - Oita University hospital, Yufu

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: After the end of the study

REFERENCES:
- [Derived] Mouri A, Kagamu H, Tamada K, Nishio M, Akamatsu H, Goto Y, Hayashi H, Miura S, Gemma A, Yoshino I, Misumi T, Saito R, Yanagitani N, Masaki F, Nokihara H, Nishino K, Seike M, Hase T, Hataji O, Takeoka H, Kawashima Y, Kuroki H, Sugimoto M, Kuriki H, Mitsudomi T. Analysis of Peripheral T Cell Profiling and Plasma Proteomics in Advanced NSCLC Patients Treated With Atezolizumab. Cancer Sci. 2026 Feb 2. doi: 10.1111/cas.70310. Online ahead of print. PMID 41627979